CLINICAL TRIAL: NCT02056964
Title: The HEART Pathway: Bridging the Gap Between Operations, Research, and Education
Brief Title: HEART Pathway Implementation
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Association of American Medical Colleges (Other); Donaghue Medical Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00025114
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Chest Pain; Acute Coronary Syndrome; Chest Pain Atypical Syndrome; Chest Pain Rule Out Myocardial Infarction
Keywords: Acute Coronary Syndrome; Chest Pain; Risk Stratification; Clinical Decision Aid; Emergency Department; Low Risk Chest Pain; Non Cardiac Chest Pain
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-HEART Pathway Implementation: Data will be collected on patients presenting to the Emergency Department (ED) with chest pain after implementation of the HEART Pathway decision aid.
- Pre-HEART Pathway Implementation: Data will be collected on patients presenting to the Emergency Department (ED) with chest pain prior to Implementation of the HEART Pathway decision aid.

SUMMARY:
The purpose of this study is to determine the effectiveness of the HEART Pathway, a clinical decision aid for the care of patients with chest pain, in a "real-world" clinical setting. This will be accomplished through the building of a transformative collaboration between research, education, and health systems operations to more effectively and efficiently provide patient care.

DETAILED DESCRIPTION:
Millions of patients with chest pain are seen in Emergency Departments (EDs) every year. Over half of ED patients with chest pain are admitted to the hospital to undergo further testing. Despite high testing rates, less than 1 in 10 patients with chest pain are ultimately diagnosed with an acute coronary syndrome (ACS) at estimated annual cost of $13 billion. Current care patterns for acute chest pain fail to focus health system resources, such as hospitalization and cardiac testing, on patients most likely to benefit.

The HEART Pathway, which combines a clinical decision aid, with two serial troponin measurements, has been developed to identify patients with chest pain who can safely be discharged without objective cardiac testing (stress testing or angiography). Prior retrospective and observational studies have established that use of the HEART Pathway reduces cardiac testing by >20%, while maintaining an acceptably low adverse event rate. We now seek to integrate the HEART Pathway into "real-world" clinical settings to determine effectiveness.

The goal of this proposal is to build a transformative collaboration bridging the gap between research, education, and health systems operations to more effectively and efficiently provide patient care. The vanguard for this collaboration seeks to improve quality of care for patients with acute chest pain by integrating the HEART Pathway into cardiovascular care delivery at Wake Forest Baptist Health (WFBH). This project will build on our prior work and provide a model for using the education and operational strengths of US academic medical centers to disseminate initiatives to improve care delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 21 years of age at the time of Emergency Department (ED) visit
* Chest discomfort consistent with possible Acute Coronary Syndrome (ACS) as indicated by the treating physician obtaining an Electrocardiogram (ECG) and cardiac biomarkers for the patient's evaluation.

Exclusion Criteria:

* New ST-segment elevation in contiguous leads on any electrocardiogram (>/= 1 mV)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is adult patients with acute chest pain, but without obvious Acute Coronary Syndrome (ACS) on Electrocardiogram (ECG). Therefore, adult patients (>21 years old) with acute chest pain, for whom the provider orders troponins, and without evidence of an ST-segment elevation myocardial infarction (STEMI) on ECG, will be included. Based on STEMI rates at Wake Forest Baptist Medical Center (WFBMC) we expect less than 5% of patients with acute chest pain to be excluded due to ECG criteria.
Sampling Method: Probability Sample
Enrollment: 14717 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Hospitalization rate | 30 Days after Emergency Department Visit

CONTACTS AND LOCATIONS:
Overall Officials: Simon A Mahler, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Rosamond W, Flegal K, Friday G, Furie K, Go A, Greenlund K, Haase N, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell CJ, Roger V, Rumsfeld J, Sorlie P, Steinberger J, Thom T, Wasserthiel-Smoller S, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2007 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2007 Feb 6;115(5):e69-171. doi: 10.1161/CIRCULATIONAHA.106.179918. Epub 2006 Dec 28. No abstract available. PMID 17194875
- [Background] McCaig LF, Nawar EW. National Hospital Ambulatory Medical Care Survey: 2004 emergency department summary. Adv Data. 2006 Jun 23;(372):1-29. PMID 16841785
- [Background] Owens PL, Barrett ML, Gibson TB, Andrews RM, Weinick RM, Mutter RL. Emergency department care in the United States: a profile of national data sources. Ann Emerg Med. 2010 Aug;56(2):150-65. doi: 10.1016/j.annemergmed.2009.11.022. Epub 2010 Jan 15. PMID 20074834
- [Background] Pope JH, Aufderheide TP, Ruthazer R, Woolard RH, Feldman JA, Beshansky JR, Griffith JL, Selker HP. Missed diagnoses of acute cardiac ischemia in the emergency department. N Engl J Med. 2000 Apr 20;342(16):1163-70. doi: 10.1056/NEJM200004203421603. PMID 10770981
- [Background] Pines JM, Isserman JA, Szyld D, Dean AJ, McCusker CM, Hollander JE. The effect of physician risk tolerance and the presence of an observation unit on decision making for ED patients with chest pain. Am J Emerg Med. 2010 Sep;28(7):771-9. doi: 10.1016/j.ajem.2009.03.019. Epub 2010 Feb 25. PMID 20837253
- [Background] Fleischmann KE, Goldman L, Johnson PA, Krasuski RA, Bohan JS, Hartley LH, Lee TH. Critical pathways for patients with acute chest pain at low risk. J Thromb Thrombolysis. 2002 Apr;13(2):89-96. doi: 10.1023/a:1016246814235. PMID 12101386
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056
- [Background] Goldstein JA, Gallagher MJ, O'Neill WW, Ross MA, O'Neil BJ, Raff GL. A randomized controlled trial of multi-slice coronary computed tomography for evaluation of acute chest pain. J Am Coll Cardiol. 2007 Feb 27;49(8):863-71. doi: 10.1016/j.jacc.2006.08.064. Epub 2007 Feb 12. PMID 17320744
- [Background] Farkouh ME, Smars PA, Reeder GS, Zinsmeister AR, Evans RW, Meloy TD, Kopecky SL, Allen M, Allison TG, Gibbons RJ, Gabriel SE. A clinical trial of a chest-pain observation unit for patients with unstable angina. Chest Pain Evaluation in the Emergency Room (CHEER) Investigators. N Engl J Med. 1998 Dec 24;339(26):1882-8. doi: 10.1056/NEJM199812243392603. PMID 9862943
- [Background] Heller GV, Stowers SA, Hendel RC, Herman SD, Daher E, Ahlberg AW, Baron JM, Mendes de Leon CF, Rizzo JA, Wackers FJ. Clinical value of acute rest technetium-99m tetrofosmin tomographic myocardial perfusion imaging in patients with acute chest pain and nondiagnostic electrocardiograms. J Am Coll Cardiol. 1998 Apr;31(5):1011-7. doi: 10.1016/s0735-1097(98)00057-6. PMID 9562001
- [Background] Sprivulis PC, Da Silva JA, Jacobs IG, Frazer AR, Jelinek GA. The association between hospital overcrowding and mortality among patients admitted via Western Australian emergency departments. Med J Aust. 2006 Mar 6;184(5):208-12. doi: 10.5694/j.1326-5377.2006.tb00416.x. PMID 16515429
- [Background] Miro O, Antonio MT, Jimenez S, De Dios A, Sanchez M, Borras A, Milla J. Decreased health care quality associated with emergency department overcrowding. Eur J Emerg Med. 1999 Jun;6(2):105-7. doi: 10.1097/00063110-199906000-00003. PMID 10461551
- [Background] Braunwald E, Antman EM, Beasley JW, Califf RM, Cheitlin MD, Hochman JS, Jones RH, Kereiakes D, Kupersmith J, Levin TN, Pepine CJ, Schaeffer JW, Smith EE 3rd, Steward DE, Theroux P, Gibbons RJ, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Smith SC Jr; American College of Cardiology; American Heart Association. Committee on the Management of Patients With Unstable Angina. ACC/AHA 2002 guideline update for the management of patients with unstable angina and non-ST-segment elevation myocardial infarction--summary article: a report of the American College of Cardiology/American Heart Association task force on practice guidelines (Committee on the Management of Patients With Unstable Angina). J Am Coll Cardiol. 2002 Oct 2;40(7):1366-74. doi: 10.1016/s0735-1097(02)02336-7. No abstract available. PMID 12383588
- [Background] Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Halperin JL, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non-ST-Elevation Myocardial Infarction); American College of Emergency Physicians; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; American Association of Cardiovascular and Pulmonary Rehabilitation; Society for Academic Emergency Medicine. ACC/AHA 2007 guidelines for the management of patients with unstable angina/non-ST-Elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non-ST-Elevation Myocardial Infarction) developed in collaboration with the American College of Emergency Physicians, the Society for Cardiovascular Angiography and Interventions, and the Society of Thoracic Surgeons endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation and the Society for Academic Emergency Medicine. J Am Coll Cardiol. 2007 Aug 14;50(7):e1-e157. doi: 10.1016/j.jacc.2007.02.013. No abstract available. PMID 17692738
- [Background] Ellestad MH, Savitz S, Bergdall D, Teske J. The false positive stress test. Multivariate analysis of 215 subjects with hemodynamic, angiographic and clinical data. Am J Cardiol. 1977 Nov;40(5):681-5. doi: 10.1016/0002-9149(77)90182-5. No abstract available. PMID 920605
- [Background] Bamberg F, Abbara S, Schlett CL, Cury RC, Truong QA, Rogers IS, Nagurney JT, Brady TJ, Hoffmann U. Predictors of image quality of coronary computed tomography in the acute care setting of patients with chest pain. Eur J Radiol. 2010 Apr;74(1):182-8. doi: 10.1016/j.ejrad.2009.03.001. Epub 2009 Apr 5. PMID 19346094
- [Background] Iskandrian AS, Heo J. Appraisal of false positive results in nuclear cardiac imaging. Am Heart J. 1990 Mar;119(3 Pt 1):708-9. doi: 10.1016/s0002-8703(05)80309-6. No abstract available. PMID 2309622
- [Background] Bach DS, Muller DW, Gros BJ, Armstrong WF. False positive dobutamine stress echocardiograms: characterization of clinical, echocardiographic and angiographic findings. J Am Coll Cardiol. 1994 Oct;24(4):928-33. doi: 10.1016/0735-1097(94)90851-6. PMID 7930226
- [Background] Einstein AJ, Henzlova MJ, Rajagopalan S. Estimating risk of cancer associated with radiation exposure from 64-slice computed tomography coronary angiography. JAMA. 2007 Jul 18;298(3):317-23. doi: 10.1001/jama.298.3.317. PMID 17635892
- [Background] Thompson RC, Cullom SJ. Issues regarding radiation dosage of cardiac nuclear and radiography procedures. J Nucl Cardiol. 2006 Jan-Feb;13(1):19-23. doi: 10.1016/j.nuclcard.2005.11.004. No abstract available. PMID 16464713
- [Background] Wagner EH. Chronic disease management: what will it take to improve care for chronic illness? Eff Clin Pract. 1998 Aug-Sep;1(1):2-4. No abstract available. PMID 10345255
- [Background] Six AJ, Backus BE, Kelder JC. Chest pain in the emergency room: value of the HEART score. Neth Heart J. 2008 Jun;16(6):191-6. doi: 10.1007/BF03086144. PMID 18665203
- [Background] Backus BE, Six AJ, Kelder JC, Mast TP, van den Akker F, Mast EG, Monnink SH, van Tooren RM, Doevendans PA. Chest pain in the emergency room: a multicenter validation of the HEART Score. Crit Pathw Cardiol. 2010 Sep;9(3):164-9. doi: 10.1097/HPC.0b013e3181ec36d8. PMID 20802272
- [Background] Backus BE, Six AJ, Kelder JC, Bosschaert MA, Mast EG, Mosterd A, Veldkamp RF, Wardeh AJ, Tio R, Braam R, Monnink SH, van Tooren R, Mast TP, van den Akker F, Cramer MJ, Poldervaart JM, Hoes AW, Doevendans PA. A prospective validation of the HEART score for chest pain patients at the emergency department. Int J Cardiol. 2013 Oct 3;168(3):2153-8. doi: 10.1016/j.ijcard.2013.01.255. Epub 2013 Mar 7. PMID 23465250
- [Background] Mahler SA, Hiestand BC, Goff DC Jr, Hoekstra JW, Miller CD. Can the HEART score safely reduce stress testing and cardiac imaging in patients at low risk for major adverse cardiac events? Crit Pathw Cardiol. 2011 Sep;10(3):128-33. doi: 10.1097/HPC.0b013e3182315a85. PMID 21989033
- [Background] Diercks DB, Peacock WF 4th, Hollander JE, Singer AJ, Birkhahn R, Shapiro N, Glynn T, Nowack R, Safdar B, Miller CD, Lewandrowski E, Nagurney JT. Diagnostic accuracy of a point-of-care troponin I assay for acute myocardial infarction within 3 hours after presentation in early presenters to the emergency department with chest pain. Am Heart J. 2012 Jan;163(1):74-80.e4. doi: 10.1016/j.ahj.2011.09.028. PMID 22172439
- [Background] Mahler SA, Miller CD, Hollander JE, Nagurney JT, Birkhahn R, Singer AJ, Shapiro NI, Glynn T, Nowak R, Safdar B, Peberdy M, Counselman FL, Chandra A, Kosowsky J, Neuenschwander J, Schrock JW, Plantholt S, Diercks DB, Peacock WF. Identifying patients for early discharge: performance of decision rules among patients with acute chest pain. Int J Cardiol. 2013 Sep 30;168(2):795-802. doi: 10.1016/j.ijcard.2012.10.010. Epub 2012 Oct 30. PMID 23117012
- [Background] Miller CD, Hwang W, Hoekstra JW, Case D, Lefebvre C, Blumstein H, Hiestand B, Diercks DB, Hamilton CA, Harper EN, Hundley WG. Stress cardiac magnetic resonance imaging with observation unit care reduces cost for patients with emergent chest pain: a randomized trial. Ann Emerg Med. 2010 Sep;56(3):209-219.e2. doi: 10.1016/j.annemergmed.2010.04.009. Epub 2010 May 31. PMID 20554078
- [Background] Hollander JE, Blomkalns AL, Brogan GX, Diercks DB, Field JM, Garvey JL, Gibler WB, Henry TD, Hoekstra JW, Holroyd BR, Hong Y, Kirk JD, O'Neil BJ, Jackson RE; Multidisciplinary Standardized Reporting Criteria Task Force. Standardized reporting guidelines for studies evaluating risk stratification of ED patients with potential acute coronary syndromes. Acad Emerg Med. 2004 Dec;11(12):1331-40. doi: 10.1197/j.aem.2004.08.033. No abstract available. PMID 15576525
- [Background] Wright RS, Anderson JL, Adams CD, Bridges CR, Casey DE Jr, Ettinger SM, Fesmire FM, Ganiats TG, Jneid H, Lincoff AM, Peterson ED, Philippides GJ, Theroux P, Wenger NK, Zidar JP, Jacobs AK. 2011 ACCF/AHA Focused Update of the Guidelines for the Management of Patients With Unstable Angina/ Non-ST-Elevation Myocardial Infarction (Updating the 2007 Guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 May 10;123(18):2022-60. doi: 10.1161/CIR.0b013e31820f2f3e. Epub 2011 Mar 28. No abstract available. PMID 21444889
- [Background] O'Connor RE, Bossaert L, Arntz HR, Brooks SC, Diercks D, Feitosa-Filho G, Nolan JP, Vanden Hoek TL, Walters DL, Wong A, Welsford M, Woolfrey K; Acute Coronary Syndrome Chapter Collaborators. Part 9: Acute coronary syndromes: 2010 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2010 Oct 19;122(16 Suppl 2):S422-65. doi: 10.1161/CIRCULATIONAHA.110.985549. No abstract available. PMID 20956257
- [Background] Miller CD, Hwang W, Case D, Hoekstra JW, Lefebvre C, Blumstein H, Hamilton CA, Harper EN, Hundley WG. Stress CMR imaging observation unit in the emergency department reduces 1-year medical care costs in patients with acute chest pain: a randomized study for comparison with inpatient care. JACC Cardiovasc Imaging. 2011 Aug;4(8):862-70. doi: 10.1016/j.jcmg.2011.04.016. PMID 21835378
- [Background] Glasgow RE, Orleans CT, Wagner EH. Does the chronic care model serve also as a template for improving prevention? Milbank Q. 2001;79(4):579-612, iv-v. doi: 10.1111/1468-0009.00222. PMID 11789118
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness: the chronic care model, Part 2. JAMA. 2002 Oct 16;288(15):1909-14. doi: 10.1001/jama.288.15.1909. PMID 12377092
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- [Derived] Ashburn NP, Snavely AC, Paradee BE, O'Neill JC, Stopyra JP, Mahler SA. Age differences in the safety and effectiveness of the HEART Pathway accelerated diagnostic protocol for acute chest pain. J Am Geriatr Soc. 2022 Aug;70(8):2246-2257. doi: 10.1111/jgs.17777. Epub 2022 Apr 5. PMID 35383887
- [Derived] Husain I, Mahler SA, Hiestand BC, Miller CD, Stopyra JP. The Impact of Accelerated Diagnostic Protocol Implementation on Chest Pain Observation Unit Utilization. Crit Pathw Cardiol. 2022 Mar 1;21(1):7-10. doi: 10.1097/HPC.0000000000000254. PMID 33534506
- [Derived] Smith LM, Ashburn NP, Snavely AC, Stopyra JP, Lenoir KM, Wells BJ, Hiestand BC, Herrington DM, Miller CD, Mahler SA. Identification of very low-risk acute chest pain patients without troponin testing. Emerg Med J. 2020 Nov;37(11):690-695. doi: 10.1136/emermed-2020-209698. Epub 2020 Aug 4. PMID 32753395
- [Derived] Stopyra J, Snavely AC, Hiestand B, Wells BJ, Lenoir KM, Herrington D, Hendley N, Ashburn NP, Miller CD, Mahler SA. Comparison of accelerated diagnostic pathways for acute chest pain risk stratification. Heart. 2020 Jul;106(13):977-984. doi: 10.1136/heartjnl-2019-316426. Epub 2020 Apr 8. PMID 32269131
- [Derived] Mahler SA, Lenoir KM, Wells BJ, Burke GL, Duncan PW, Case LD, Herrington DM, Diaz-Garelli JF, Futrell WM, Hiestand BC, Miller CD. Safely Identifying Emergency Department Patients With Acute Chest Pain for Early Discharge. Circulation. 2018 Nov 27;138(22):2456-2468. doi: 10.1161/CIRCULATIONAHA.118.036528. PMID 30571347
- [Derived] Mahler SA, Burke GL, Duncan PW, Case LD, Herrington DM, Riley RF, Wells BJ, Hiestand BC, Miller CD. HEART Pathway Accelerated Diagnostic Protocol Implementation: Prospective Pre-Post Interrupted Time Series Design and Methods. JMIR Res Protoc. 2016 Jan 22;5(1):e10. doi: 10.2196/resprot.4802. PMID 26800789
- See also: Wake Forest Baptist Medical Center — http://www.wakehealth.edu